CLINICAL TRIAL: NCT07374510
Title: An Open-Label Combined Randomized, Blinded, Placebo- and Active-Controlled Phase Ia Clinical Trial: Evaluate the Safety and Immunogenicity of the Group ACYW135X Meningococcal Conjugate Vaccine in Individuals Aged 2 to 59 Years
Brief Title: Phase Ia Clinical Trial of Group ACYW135X Meningococcal Conjugate Vaccine
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-ACYWX-1001
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Meningococcal Meningitis
Keywords: ACYW135X; vaccine; phase 1
MeSH Terms: conditions — Meningitis, Meningococcal | interventions — CRM197 (non-toxic variant of diphtheria toxin)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- high-dose experimental group (Experimental): 2~59 years old
  Interventions: Biological: high-dose Group ACYW135X Meningococcal Conjugate Vaccine
- medium-dose experimental group (Experimental): 2~59 years old
  Interventions: Biological: medium-dose Group ACYW135X Meningococcal Conjugate Vaccine
- low-dose experimental group (Experimental): 2~6 years old
  Interventions: Biological: low-dose Group ACYW135X Meningococcal Conjugate Vaccine
- placebo group (Placebo Comparator): 2~6 years old
  Interventions: Biological: Placebo
- active control group (Active Comparator): 2~3 years old
  Interventions: Biological: Group ACYW135 Meningococcal Conjugate Vaccine (CRM197)

INTERVENTIONS:
Biological: high-dose Group ACYW135X Meningococcal Conjugate Vaccine — high-dose Group ACYW135X Meningococcal Conjugate Vaccine
  Arms: high-dose experimental group
Biological: medium-dose Group ACYW135X Meningococcal Conjugate Vaccine — medium-dose Group ACYW135X Meningococcal Conjugate Vaccine
  Arms: medium-dose experimental group
Biological: low-dose Group ACYW135X Meningococcal Conjugate Vaccine — low-dose Group ACYW135X Meningococcal Conjugate Vaccine
  Arms: low-dose experimental group
Biological: Group ACYW135 Meningococcal Conjugate Vaccine (CRM197) — Group ACYW135 Meningococcal Conjugate Vaccine (CRM197)
  Other Names: Menhycia
  Arms: active control group
Biological: Placebo — placebo
  Arms: placebo group

SUMMARY:
This trial adopts an open-label design combined with randomized, blinded, placebo-controlled and active-controlled design. The purpose of this trial is to evaluate the safety and immunogenicity of a Group ACYW135X Meningococcal Conjugate Vaccine. This study is planned to enroll 150 participants in total, with healthy individuals aged 2 to 59 years as participants. Among them, participants aged 18 to 59 years and 7 to 17 years will be assigned to the open-label design arm, while participants aged 4 to 6 years will be assigned to the randomized, blinded, placebo-controlled design arms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged 2 to 59 years;
* The participant and/or their legal guardian can understand and voluntarily sign the informed consent form (for participants aged 8 to 17 years, the form must be signed jointly by the participant and their legal guardian);
* Be willing and able to comply with all visit schedules, sample collection procedures, vaccination protocols and other trial-related requirements, and maintain contact at any time during the study period;
* Provide valid legal identification documents of the participant and/or their legal guardian;
* Participants of childbearing potential and their sexual partners shall voluntarily adopt effective contraceptive measures from the date of signing the informed consent form until 3 months after the administration of the investigational vaccine, with no plans for sperm or egg donation during this period.

Exclusion Criteria:

* History of meningococcal disease;
* History of asthma; history of hypersensitivity to any vaccine or vaccine components (including serogroup A/C/Y/W135/X meningococcal capsular polysaccharide, mannitol, sucrose, disodium hydrogen phosphate, sodium dihydrogen phosphate, sodium chloride, and water for injection), manifested as symptoms such as urticaria, dyspnea, or angioedema; or history of other severe adverse reactions following previous vaccination;
* For children aged 2 to 6 years: history of previous vaccination with group ACYW135 meningococcal polysaccharide vaccine; or history of previous vaccination with any meningococcal conjugate vaccine other than group AC meningococcal conjugate vaccine; an interval of ≤ 12 months from the last dose of group A or group AC meningococcal polysaccharide vaccine or group AC meningococcal conjugate vaccine; history of vaccination with meningococcal conjugate vaccine since reaching 1 year of age. No vaccination history restrictions apply to participants aged 7 to 59 years;
* Presence of autoimmune diseases or immunodeficiency diseases (including but not limited to systemic lupus erythematosus, ankylosing spondylitis, autoimmune thyroid diseases, asplenia, functional asplenia, and HIV infection);
* Presence of coagulation disorders (e.g., coagulation factor deficiency, thrombocytopathy), or a history of significant bleeding, hematoma, or ecchymosis following previous intramuscular injection or venipuncture;
* History of severe diseases or current diagnosis of severe chronic diseases (including but not limited to severe cardiovascular diseases, uncontrolled hypertension, hematological diseases, hepatic and renal diseases, gastrointestinal diseases, respiratory diseases, malignant tumors, and history of major organ transplantation);
* Presence of severe congenital malformations, genetic defects, or malnutrition;
* Presence or history of severe neurological diseases (epilepsy, convulsions, or seizures) or psychiatric disorders, or a family history of psychiatric disorders;
* Chronic alcohol abuse [weekly alcohol consumption > 14 standard drinks (1 standard drink = 14 grams of 100% alcohol ≈ 360 mL beer, 150 mL wine, or 45 mL distilled spirits/liquor)] or a history of substance abuse (repeated and excessive use of narcotic drugs, psychotropic drugs, volatile organic solvents, etc.);
* Receipt of immunosuppressive therapy or other immunomodulatory therapy for ≥ 14 days within the past 6 months (prednisone ≥ 20 mg/day or ≥ 2 mg/kg/day, or its equivalent dose); receipt of cytotoxic therapy; or planned receipt of such therapies during the study period;
* Receipt of blood products within 3 months prior to the administration of the investigational vaccine;
* Receipt of other investigational drugs or vaccines within 3 months prior to the administration of the investigational vaccine, or planned receipt of such drugs or vaccines during the study period;
* Receipt of live attenuated vaccines or nucleic acid vaccines within the past 14 days, or receipt of subunit vaccines or inactivated vaccines within the past 7 days;
* Participants who are breastfeeding, pregnant, or planning to become pregnant within 3 months after vaccination in this trial;
* Presence of any acute diseases or acute exacerbation of chronic diseases within the past 7 days, or known or suspected active infections;
* Clinically significant abnormal findings in laboratory tests：

  1. Hematological parameters: white blood cell count, hemoglobin, platelet count;
  2. Biochemical parameters: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), blood glucose;
  3. Urinalysis parameters: urine protein (PRO);
* Axillary temperature > 37.0℃ prior to vaccination, or other vital sign measurements beyond the reference range;
* Presence of skin damage, inflammation, ulceration, rash, or scarring at the intended injection site that may interfere with vaccination or observation of local reactions;
* Any other factors that, in the investigator's judgment, render the participant unsuitable for participation in this clinical trial.

Ages: 2 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of experimental vaccine among participants in different age groups (based on adverse reactions) | 30 days
  The incidence rates of adverse reactions 30 days after vaccination

SECONDARY OUTCOMES:
Evaluate the safety of experimental vaccine among participants in different age groups (based on AE and laboratory abnormalities) | 30 days
  The incidence rate of adverse events 30 days after vaccination
Evaluate the safety of experimental vaccine among participants in different age groups (based on AE and laboratory abnormalities) | 3 days
  The incidence rate of clinically significant abnormal blood biochemistry, blood routine, and urine routine indexes within 3 days after vaccination
Evaluate the safety of experimental vaccine among participants in different age groups (based on AE and laboratory abnormalities) | 6 months
  The incidence rate of serious adverse events 6 months after vaccination
Evaluate the immunogenicity of experimental vaccine among participants aged 2~6 years old | 30 days
  The seropositive rates, seroconversion rate, GMT and GMFR of Nm antibody against serogroups A, C, Y, W135, and X at 30 days after vaccination
Evaluate the immunogenicity of experimental vaccine among participants aged 2~6 years old | 30 days
  The proportion of Nm antibody against serogroups A, C, Y, W135, and X with titer ≥ 1:16, ≥ 1:32, ≥ 1:64, and ≥ 1:128 at 30 days after vaccination